CLINICAL TRIAL: NCT01081444
Title: Effect of Pharyngeal Inhibition Induced by Repetitive Transcranial Stimulation in Post Stroke Dysphagia
Brief Title: Repetitive Transcranial Stimulation (rTMS) in Post Stroke Dysphagia
Acronym: rTMS AVC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007/122/HP
Record Dates: First submitted 2009-08-14; First posted 2010-03-05 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Dysphagia; Stroke
Keywords: repetitive transcranial stimulation
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Active rTMS
  Interventions: Device: rTMS
- 2 (Placebo Comparator): sham rTMS
  Interventions: Device: Placebo rTMS

INTERVENTIONS:
Device: rTMS — effective and active cortical magnetic stimulations
  Arms: 1
Device: Placebo rTMS — non active cortical magnetic stimulation
  Arms: 2

SUMMARY:
The aim of this study is to assess if rTMS on healthy hemisphere at one hertz could improve patients with post stroke dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* dysphagia
* first episode of stroke

Exclusion Criteria:

* swallowing disorder before stroke
* previous episode of stroke
* MMS < 20 no consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Videofluoroscopy and high resolution manometry | day 0, day 14, day 30, day45

CONTACTS AND LOCATIONS:
Overall Officials: Eric VERIN, MD-PhD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Physiology, Rouen University Hospital, Rouen, France